# Statistical Analysis Plan: Mock-up Tables and Figures

Version 1.0, 25-JAN-2022

**Protocol Number: CX4945-AV01-IIT** 

A Phase II, Randomized and Controlled Investigator Initiated Trial Evaluating Safety, Pharmacokinetics and Clinical Benefit of Silmitasertib (CX-4945) in Outpatient Adult Subjects with Moderate Coronavirus Disease 2019 (COVID-19)

Protocol version: Amendment 1.0, 11MAY2021 Sponsor-Investigator: Dr. Chris Recknor, MD Drug Provider: Senhwa Biosciences, Inc.



#### **Table of Contents**

| Statisti | ical Analysis Plan: Mock-up Tables and Figures | 1 |
|---|---|---|
| Table o | of Contents | 2 |
| 1 St | Statistical Changes from Study Protocol | 3 |
| 1.1 | Visit Adjustment | |
| 1.2 | Per-Protocol (PP) Population | |
| 1.3 | Treatment Compliance of CX-4945 | 3 |
| 1.4 | Analysis Method | |
| | .4.1 Inferential Statistics | |
| | .4.3 Method for Continuous Data | |
| | .4.4 Method for Categorical Data | |
| 1.5 | Method for Handling Missing Value | 5 |
| 1.6 | Pharmacokinetics Analyses | 5 |
| 2 P | Protocol Versions and Protocol Amendments | 6 |
| 3 M | Mock-up Tables and Figures | 7 |
| 3.1 | Analysis of Continuous Data | 7 |
| 3.2 | Analysis of Categorical Data | 7 |
| Instruc | ctions and Abbreviations: | 8 |
| 14 T | TABLES and FIGURES | 11 |
| 14.1 | DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS | 12 |
| 14 | 4.1.1 Screen Failures and Subject Disposition by Study Site | 12 |
| | 4.1.2 Study Termination, Subject Disposition and Protocol Deviation | |
| | 4.1.3 Study Visits | |
| | 4.1.4 Demographic Data | |
| | 4.1.5 Cotoliavitus Disease 2019 (COVID-19) History 4.1.6 General Medical History and Concurrent Disease/Status | |
| | 4.1.7 Concomitant Medications | |
| | 4.1.8 Best Supportive / Standard Of Care Procedures | |
| | 4.1.9 Study Drug Administration, Compliance and Exposure | |
| 14.2 | | |
| | 4.2.1 COVID-19-Related Clinical Signs | |
| _ | 4.2.2 Covid-19-Related Symptoms | |
| | 4.2.3 Nasopharyngeal Swab RT-PCR Result and SARS-COV-2 Viral Load | |
| | 4.2.4 Clinical Status - NIAID 8-Point Clinical Progression Outcomes Scale | |
| | 4.2.5 EQ-5D-5L | |
| 14.3 | S SAFETY DATA | 25 |
| 14 | 4.3.1 Treatment Emergent Adverse Event – Subject Based Analyses | 25 |
| 14 | 4.3.2 Laboratory Examination – Hematology | 28 |
| | 4.3.3 Laboratory Examination – Chemistry | |
| | 4.3.4 Laboratory Examination – Inflammatory Marker | |
| | 4.3.5 Laboratory Examination – Coagulation | |
| | 4.3.6 Laboratory Examination – Urinalysis | |
| | 4.3.7 Physical Examination | |
| | 4.3.8 Vital Signs, Body Weight and SpO2 | |
| 14 | 7.5.7 Electrocatulogram (ECO) | |



#### 1 Statistical Changes from Study Protocol

The statistical analysis methods will follow study protocol version amendment 1.0 (11-MAY-2021, exceptions and clarifications are described below:

#### 1.1 Visit Adjustment

Visit 6 is End of Treatment (EOT) Visit, Treatment Discontinuation Visit or Early Withdrawal Visit at/before EOT. Data of visit 6 not in its visit window will be shifted to corresponding scheduled visit for analysis as in table below (marked '\*'). Visit name will be presented as 'Adjusted Visit' for the visits reallocated to its original scheduled visit or the next visit after preceding scheduled visit.

| | Visit 6 to Visit 3~6 |
|---|---|
| COVID-19-Related Symptoms | * |
| Clinical Status - NIAID 8-Point Clinical Progression Outcomes Scale | * |
| Laboratory Examination | * |
| Vital Signs, Pulse Oxygen Saturation (SpO2) and | * |
| COVID-19-Related Clinical Signs | ' |

#### 1.2 Per-Protocol (PP) Population

According to the protocol, subject with major protocol violation shall be excluded from PP population. The definition shall be revised to 'The PP population is defined as the set of patients who meet the ITT population requirements and are not associated with any major protocol violations *relevant to efficacy analysis*'.

#### **14.1.1.1** 9.7.1.2. Per Protocol (PP) Population

The PP population is defined as the set of patients who meet the ITT population requirements and are not associated with any major protocol violations. This population will be identified before the database lock. This population will be used as the supportive analysis population for analysis of the primary and secondary efficacy endpoints.

#### 1.3 Treatment Compliance of CX-4945

There is no definition of compliance in the protocol, it's defined as below.

| Treatment Compliance [%]= | # of times of CX-4945 actually administered | *100% |
|---|---|---|
| Treatment Compnance [70]— | (Treatment Duration) * (2 times of administration/day) | |

 $Treatment\ Duration\ [days] = the\ last\ administration\ date-the\ first\ administration+Adjustment$ 

| The first administration time | The last administration time | Adjustment |
|-------------------------------|------------------------------|------------|
| Morning | Morning | +0.5 |
| Morning | Evening | +1 |
| Evening | Morning | +0 |
| Evening | Evening | +0.5 |

#### 1.4 Analysis Method

#### 1.4.1 Inferential Statistics

According to the protocol, no inferential statistics was planned. In the SAP, the inferential testing will be done as appropriate for treatment comparison.



Silmitasertib (CX-4945) for COVID-19

#### 9.8.4. Study Outcome Assessment

For continuous variables data will be summarized by treatment using n, mean, SD, minimum and maximum values. For categorical variables data will be summarized by treatment using frequency and percentage. No inferential statistics are planned. The Safety population will be used for the analysis of safety outcomes.

#### 1.4.2 Method for Time to Event Data

The endpoints about time to event data as below table will be compared between treatment groups by using log-rank test, and corresponding response proportion will be presented by using Kaplan-Meier methods.

- Time to COVID-19-Related Clinical Signs Normalization
- Time to Oxygen Saturation Level Normalization
- Time to moderate COVID-19-Related Symptoms Resolution
- Time to SARS-COV-2 Viral Clearance
- Time to Improvement on NIAID 8-Point Clinical Progression Outcomes Scale (additional analysis, not mentioned in the protocol)
- Time to Improvement on EQ-5D-5L Imaginable Health Status (additional analysis, not mentioned in the protocol)

Considering the early censor on time to response (Normalization / Recovery / Viral Clearance / Improvement) data will result in over optimistic in statistical results, two data estimation methods below will be used for the sensitive analyses. Results will be claimed as robust if the results of both methods are consistent.

Time to Response (days), Best Case Scenario

- = Days to first response for responder,
- = Days to last observation for non-responder (censored)

Time to Response (days), Worst Case Scenario

- = Days to first response for responder,
- = Days to planned last observation date (31 for EQ-5D-5L and SARS-COV-2 Viral Clearance at visit 7, 45 for others at visit 8) for non-responder (censored)

Days to first response = date of first response – the first treatment date/time + 1Days to last observation = date of last evaluation – the first treatment date/time + 1For Arm SOC, the first treatment date is the date of visit 2

#### 1.4.3 Method for Continuous Data

Demographics, baseline characteristics and continuous efficacy data will be analyzed by using two sample t test or Wilcoxon rank-sum test as appropriate. Net changes from pre-treatment laboratory test results and vital signs will be analyzed by using ANCOVA model with baseline value as covariate or Wilcoxon rank-sum test as appropriate.

#### 1.4.4 Method for Categorical Data

Categorical data will be analyzed by using the Fisher's exact test or Chi-square test as



appropriate. Ordinal data will be analyzed by using Mantel-Haenszel chi-square test on given scores.

#### 1.5 Method for Handling Missing Value

According to protocol, multiple imputation methods were planned to be done for efficacy evaluations using PROC MI of SAS. Since the sample size is relative small for both treatments, predictive model for multiple imputation is not realistic. Additional statistics on LOCF (Last Observation Carry Forward) data will be presented for by-visit efficacy analysis.

#### 9.7.3. Missing Data

The method for handling missing data will be included in the statistical analysis plan. Every effort will be made to obtain required data at each scheduled evaluation from all patients who have been randomized in the study to minimize missing data. However, in the event when there are missing data the following imputation methods will be used. For efficacy evaluations, multiple imputation methods will be used to handle missing data and will be detailed in the SAP. This imputation method is a robust method to impute potential missing measurements. The imputation will be carried out in SAS version 9.4 or later using PROC MI.

#### 1.6 Pharmacokinetics Analyses

Pharmacokinetics data will not be provided, and PK parameters will not be analyzed per sponsor's decision, and therefore it is not covered in the SAP.



#### 2 Protocol Versions and Protocol Amendments

The first subject was enrolled on 3-Dec-2020, and the last subject is expected to be dismissed on 7-Oct-2021. All applied protocol and CRF versions are listed as below.

| No. | <b>Protocol Version</b> | CRF Version | IRB Approval | FDA Approval |
|---|---|---|---|---|
| 1 | 3.0, 20OCT2020 | 1.1, 12OCT2021 | 5-Nov-2020 | 3-Nov-2020 |
| 2 | Amendment 1.0,<br>11MAY2021 | 1.0, 06SEP2021 | 24-May-2021 | 24-Jun-2021 |



#### 3 Mock-up Tables and Figures

The Mock-up "TABLES and FIGURES" is planned according to ICH E3, in which relevant Clinical Study Report (CSR) section is 14. The words shadowed below are to be adjusted or repeated upon real data, or just for notification.

#### 3.1 Analysis of Continuous Data

For ANOVA / ANCOVA / T test (two sample t test) noted in the mock-up table, Wilcox\_t (Wilcoxon rank-sum test in t approximation) will be applied if normality assumption is not valid (p-value of Shapiro-Wilk normality test  $\leq 0.05$ ).

#### 3.2 Analysis of Categorical Data

C/F noted in the mock-up table, Chi-Square test is applied when no cell have expected count < 1 and <=20% of the cells are with expected count < 5, otherwise Fisher's exact test will be applied.



Silmitasertib (CX-4945) for COVID-19

#### **Instructions and Abbreviations:**

#### (1) Site ID <u>CCC</u>::

| Site ID | Site Name | Site Code |
|---------|------------------------------------------|-----------|
| 001 | Center for Advanced Research & Education | CARE |
| 002 | CA' Research | CAR |

#### (2) Treatment Group:

CX-4945: The best supportive / standard of care + CX-4945 1000 mg BID,

SOC: The best supportive / standard of care

#### (3) Population

• ITT (Intention-To-Treat):

All randomized patients

Safety Population:

Receiving at least one dose of CX-4945 or being randomized to the standard of care arm.

• PP (Per-Protocol):

A subset of ITT and Safety population who are not associated major protocol deviation relevant to efficacy analysis.

If Safety Population and ITT are the same, these two populations will be combined as 'Safety Population and Intention-To-Treat' if results of both populations are to be presented in the same table.

(4) For Visit Name (in Tables and Figures) and Visit Code (in Subject Data Listing):

| Visit No. | Visit Description | Visit Day | Visit Name | Visit Code |
|---|---|---|---|---|
| 1 | Screening Visit | <b>-</b> 7 ∼ <b>-</b> 1 | Visit 1 (Screening) | V01 |
| 2 | Treatment Visit (Day 1) | 1 | Visit 2 (Day 1) | V02D01T |
| 3 | Treatment Visit (Day 4) | 4 ± 1 | Visit 3 (Day 4) | V03D04T |
| 4 | Treatment Visit (Day 8) | 8 ± 1 | Visit 4 (Day 8) | V04D08T |
| 5 | Treatment Visit (Day 11) | 11 ± 1 | Visit 5 (Day 11) | V05D11T |
| 6 | End of Treatment (EOT)Visit (Day 14) | 14 ± 1 | Visit 6 (Day 14, EOT) | V06D14E |
| 7 | Follow-up 1 Visit (Day 28) | $28 \pm 3$ | Visit 7 (Day 28, F1) | V07D28F |
| 8 | Follow-up 2 Visit (Day 45) | 45 ± 3 | Visit 8 (Day 45, F2) | V08D45F |
| 9 | Follow-up 3 Visit (Day 60) | 60 ± 3 | Visit 9 (Day 60, F3) | V09D60F |
| | Unscheduled Visit | - | - | UV |

#### (5) Efficacy Endpoints:

#### • Time to COVID-19-Related Clinical Signs Normalization: Normal when all below are met

- (1) Fever is <36.6°C from axillary site, or < 37.2°C from oral site, or < 37.8°C from rectal or tympanic site, or <37.2°C from forehead by using non-contact infrared thermometers
- (2) Respiratory rate is < 20 bpm while breathing room air
- (3) SpO2  $\geq$  96% in room air without shortness of breath or dyspnea caused by COVID-19
- (4) Heart rate < 90 beats per minute

If some signs listed above were caused by other conditions documented in the medical history and started before COVID-19, the patient can be considered as recovered, when these signs return to the previous (pre-COVID-19) values

• Oxygen Saturation Level Normalization: Normal when SpO2  $\geq$  96%

#### • Resolution of moderate COVID-19-Related Symptoms when all below are met:

- No key COVID-19-related symptoms scored higher than 1.
- If some symptoms were caused by other conditions documented in the medical history and started before COVID-19 (e.g, insomnia), the patient can be considered as recovered, when these symptoms return to the previous (pre-COVID-19) value.
- SARS-COV-2 Viral Clearance: negative RT-PCR



Silmitasertib (CX-4945) for COVID-19

#### • NIAID 8-Point Clinical Progression Outcomes Scale:

- 1 Death
- 2 Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
- 3 Hospitalized, on non-invasive ventilation or high flow oxygen devices
- 4 Hospitalized, requiring supplemental oxygen
- 5 Hospitalized, not requiring supplemental oxygen requiring ongoing medical care (COVID-19 related or otherwise)
- 6 Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care
- 7 Not hospitalized, limitation on activities and/or requiring home oxygen
- 8 Not hospitalized, no limitations on activities

# • EQ-5D-5L Imaginable Health Status Improvement: Imaginable Health Status <90 at baseline and ≥ 90 after baseline

#### • Time to Response (Normalization / Resolution / Viral Clearance / Improvement)

Time to Response (days), Best Case Scenario

- = Days to first response for responder,
- = Days to last observation for non-responder (censored)

Time to Response (days), Worst Case Scenario

- = Days to first response for responder,
- = Days to planned last observation date (31 for EQ-5D-5L and SARS-COV-2 Viral Clearance at visit 7, 45 for others at visit 8) for non-responder (censored)

Days to first response = date of first response - the first treatment date/time + 1 Days to last observation = date of last evaluation - the first treatment date/time + 1 For Arm SOC, the first treatment date is the date of visit 2

(6) For Clinical Relevance

CS: abnormal and clinically significant LLN: lower limit of normal range NCS: abnormal but not clinically significant ULN: upper limit of normal range

(7) For Transition of Clinical Relevance

Relieved CS (Medical History or Adverse Event) at baseline to Normal / NCS at

visit.

Unchanged Including Normal at baseline to NCS at visit, NCS at baseline to Normal

at visit

Worsened (Medical History) Normal / NCS at baseline to CS (Medical History) at visit

Worsened (Adverse Event) Normal / NCS / CS (Medical History) at baseline to CS (Adverse Event)

at visit

If both 'Medical History' and 'Adverse Event' are checked for 'CS', it will be counted as 'Adverse Event' only.

(8) Abbreviations of Statistics

N: number of non-missing values ANOVA: analysis of variance M: missing, not available ANCOVA: analysis of covariance

Missing: number of missing values

Mean: mean of values

CHISQ: Chi-Square test
FISHER: Fisher's exact test

SD: standard deviation of values MHCHISQ: Mantel-Haenszel chi-square test on given scores

Q1: 25% quartile of values T: two sample t test

Q3: 75% quartile of values W: Wilcoxon rank-sum test

Median: median of values Diff.: difference

IQR: inter-quartile-range (IQR=Q3-Q1)

Min: minimum of values
Max: maximum of values
CI: confidence interval
LS-mean: least-square mean

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc. Protocol No.: CX4945-AV01-IIT  A2 Healthcare Taiwan Co.



Silmitasertib (CX-4945) for COVID-19

#### For CI and p-value (WI, within group):

t denotes by using one sample t-test w denotes wilcoxon sign rank test (determined by Shapiro-Wilk normality test)

#### For CI and p-value (between groups):

Wilcox\_t denotes Wilcoxon rank-sum test (Mann-Whitney U Test) in t approximation Wilcox\_z denotes Wilcoxon rank-sum test (Mann-Whitney U Test) in z approximation ANOVA denotes Treatment effect in ANOVA model ANCOVA denotes Treatment effect in ANCOVA model For 95% CI (HL), HL denotes CI using Hodges-Lehman for median



Protocol No.: CX4945-AV01-IIT

#### **Statistical Analysis Plan: Mock-up Tables and Figures**

Silmitasertib (CX-4945) for COVID-19

#### 14 TABLES AND FIGURES

- The texts in shaded Italic are for programming note.
- Column of Study Site includes columns of {001-CARE, 002-CAR, Total}
- Column of Treatment Group includes columns of {CX-4945, SOC, Total}
- Column 'Difference' denotes pairwise comparison statistics.
- Multi-Selection means 'A subject may be counted in more than one category'
- *Description in* <...> *will be presented according to data values.*
- For column p-value: refer to Abbreviations of statistics in [Instructions and Abbreviations] above.
- For Groups Diff., SC = CX-4945, SS = SOC, T denotes two sample t test, W denotes Wilcox t (Wilcoxon rank-sum test in t approximation), C denotes Chi-Square test, F denotes Fisher's exact test

A2 Healthcare Taiwan Co.



#### 14.1 DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS

# 14.1.1 Screen Failures and Subject Disposition by Study Site Population: All Screened Subjects / Randomized Subjects

| Characteristics | Study Site |
|---------------------------------------------|--------------|
| | <u> </u> |
| . All Screened Subjects | |
| N | XXX |
| ~Randomized Subjects | XXX (XXX.X%) |
| . Population of Randomized Subjects | |
| N | XXX |
| ITT | XXX (XXX.X%) |
| ~ Safety | XXX (XXX.X%) |
| $\sim PP$ | XXX (XXX.X%) |
| ~ Non-PP | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| . Treatment Arm of Randomized Subjects | |
| N | XXX |
| CX-4945 | XXX (XXX.X%) |
| SOC | XXX (XXX.X%) |
| . Protocol Deviation of Randomized Subjects | |
| (Multi-Selection by Major/Minor & Category) | |
| N | XXX |
| ~ Any Protocol Deviation | XXX (XXX.X%) |
| ~ Major Protocol Deviation | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| ~ Minor Protocol Deviation | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| ••• | |



# 14.1.2 Study Termination, Subject Disposition and Protocol Deviation Population: Intention-to-Treat Population

| Characteristics | Treatment Group |
|----------------------------------------|--------------------|
| Study Tormination | |
| . Study Termination N | XXX |
| Study Completed | XXX (XXX.X%) |
| Study Not Completed | XXX (XXX.X%) |
| ~ Withdrew consent | XXX (XXX.X%) |
| ~ Protocol issue | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| . Study Duration [days] | TW |
| N (Missing) | $\overline{0.XXX}$ |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| . Population | |
| N | XXX |
| Safety | XXX (XXX.X%) |
| ~ PP | XXX (XXX.X%) |
| ~ Non-PP | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| . Protocol Deviation (Multi-Selection) | |
| N | XXX |
| ~ Any Protocol Deviation | XXX (XXX.X%) |
| ~ Major Protocol Deviation | XXX (XXX.X%) |
| ~ <reason 1=""></reason> | XXX (XXX.X%) |
| ~ <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| ~ Minor Protocol Deviation | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| | XXX (XXX.X%) |

Study Duration [days] = Date of Termination - Visit 1, or alternatively as the last visit date - Visit 1



#### 14.1.3 Study Visits

| Population: Inter | ntion-to-T | Treat Pop | pulation |
|-------------------|------------|-----------|----------|
|-------------------|------------|-----------|----------|

| Population: Intention-to-Treat Population | |
|---|---|
| Characteristics | Treatment Group |
| . Repeat Variable:<br>Study Visits Completed on ITT Population (Multi-Se<br>Study Visits Completed on Safety Population (Multi-<br>Study Visits Completed on PP Population (Multi-Sel | -Selection by Visit) |
| Adjusted Visits Completed on ITT Population (Multi-<br>Adjusted Visits Completed on Safety Population (Multi-<br>Adjusted Visits Completed on PP Population (Multi-<br>N | ulti-Selection by Visit) Selection by Visit) XXX |
| Visit 1 (Screening) | XXX (XXX.X%) |
| Visit 2 (Day 1) | XXX (XXX.X%) |
| Visit 3 (Day 4) ~In-Person ~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 4 (Day 8) ~In-Person ~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 5 (Day 11) ~In-Person ~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 6 (Day 14, EOT)<br>~In-Person<br>~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 7 (Day 28, F1) ~In-Person ~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 8 (Day 45, F2)<br>~In-Person<br>~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 9 (Day 60, F3)<br>~In-Person<br>~Remote (Phone/Telehealth) | XXX (XXX.X%)<br>XXX (XXX.X%)<br>XXX (XXX.X%) |



Silmitasertib (CX-4945) for COVID-19

# **14.1.4 Demographic Data** Population: Intent-to-Treat Population

| Characteristics | Treatment Group | P-value |
|---|---|---|
| . Study Site | | |
| N (Missing) | XXX (XXX) | |
| 001-CARE | XXX (XXX.X%) | |
| 002-CAR | XXX (XXX.X%) | |
| . Repeat Variable: | | |
| Age [Y/O], Baseline Body Weight [kg], Body Height [cm], | | |
| Baseline BMI [kg/m^2] | | T/W |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Mean (SD) | XXX (XXX) | |
| Median (IQR) | XXX (XXX) | |
| Q1~Q3 | XXX~XXX | |
| Min~Max | XXX~XXX | |
| . Gender | | C/F |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Male | XXX (XXX.X%) | |
| Female | XXX (XXX.X%) | |
| . Race | | |
| N (Missing) | XXX (XXX) | |
| Black /African American | XXX (XXX.X%) | |
| American Indian or Alaska Native | XXX (XXX.X%) | |
| Asian | XXX (XXX.X%) | |
| Native Hawaiian or Other Pacific Islander | XXX (XXX.X%) | |
| White | XXX (XXX.X%) | |
| . Ethnicity | | C/F |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Hispanic or Latino | XXX (XXX.X%) | |
| Not Hispanic or Latino | XXX (XXX.X%) | |

Age [years old]= (Date of informed consent obtained - birth date)/365.25 rounded down to the nearest

BMI [kg/m^2]= Weight [kg] / (Height [cm])^2 \* 10000 Baseline is Visit 2 or alternatively as Visit 1 if Visit 2 data is not available.



Silmitasertib (CX-4945) for COVID-19

#### Coronavirus Disease 2019 (COVID-19) History 14.1.5

Population: Intent-to-Treat Population

| Characteristics | Treatment Group | P-value |
|---------------------------------------------|-------------------|---------|
| . Repeat Variable: | | |
| Disease Duration [days], | | |
| Symptom Duration [days], | | |
| Symptom Duration up to Randomization [days] | | TW |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Mean (SD) | XXX (XXX) | |
| Median (IQR) | XXX (XXX) | |
| Q1~Q3 | XXX~XXX | |
| Min~Max | XXX~XXX | |
| . COVID-19 Vaccination History | | |
| N | XXX | |
| At least one below [Event#:Subj#] | XXX : XXX (XXX.X% | ) |
| ~ AstraZeneca | XXX : XXX (XXX.X% | ) |
| ~ Johnson & Johnson | XXX : XXX (XXX.X% | ) |
| ~ Pfizer | XXX : XXX (XXX.X% | ) |
| ~ Moderna | XXX : XXX (XXX.X% | ) |

Disease Duration [days] = (date of screening visit – date of first positive RT-PCR for testing COVID-19), Symptom Duration [days] = (date of screening visit – start date of COVID-19 self-reported by patient), missing day is estimated as 15, missing month is estimated as Jul-01, full unknown is missing

#### 14.1.6 **General Medical History and Concurrent Disease/Status**

Population: Intent-to-Treat Population

| Characteristics | Treatment Group |
|---------------------------------------|-----------------|
| . General Medical History | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| . Current Condition (Multi-Selection) | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| ••• | |

Current condition lists the medical histories that are ongoing or with end date  $\geq$  date of visit 2



#### 14.1.7 **Concomitant Medications**

Population: Intent-to-Treat Population / Safety Population

| Characteristics | Treatment Group |
|---|---|
| Repeat Population: <see above="" populations=""></see> | - |
| Repeat Variable: Prior Medication, Concomitant Medication | |
| (Multi-Selection by Highest ATC Level Class and ATC Preferred Term) | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| ~ < Highest ATC Level Class 1> | XXX (XXX.X%) |
| ~ <atc 1="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ <atc 2="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ < Highest ATC Level Class 2> | XXX (XXX.X%) |
| ~ <atc 1="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ <atc 2="" preferred="" term=""></atc> | XXX (XXX.X%) |

WHODrug Global B3-format September 1, 2020 is used for coding

Prior Medication: medications onset prior to Day 1

Concomitant Medication: medications applied on / after Day 1



Silmitasertib (CX-4945) for COVID-19

#### 14.1.8 Best Supportive / Standard Of Care Procedures

| opulation: Intent-to-Treat Population Characteristics | Treatment Group | P-value |
|---|---|---|
| - Repeat Duration: | | |
| Prior Procedure, Concomitant Procedure, Post Procedure | | |
| Repeat Variable: | | |
| Subject with Best Supportive / Standard Of Care Procedure | | |
| (Multi-Selection by Highest ATC Level Class and ATC Pr | referred Term) | |
| N | XXX | C/F |
| At least one below [Day#:Subj#] | XXX:XXX(XXX.X%) | 0.XXXX |
| Extracorporeal Membrane oxygenation | XXX : XXX (XXX.X%) | 0.XXXX |
| Fluid management | XXX : XXX (XXX.X%) | 0.XXXX |
| Mechanical Ventilation | XXX : XXX (XXX.X%) | 0.XXXX |
| ~ High-flow oxygen | XXX: XXX (XXX.X%) | 0.XXXX |
| ~ Supplemental oxygen | XXX : XXX (XXX.X%) | 0.XXXX |
| ~ Noninvasive ventilation | XXX : XXX (XXX.X%) | 0.XXXX |
| ~ Extracorporeal membrane oxygenation (ECMO) | XXX : XXX (XXX.X%) | 0.XXXX |
| ~ Other | XXX : XXX (XXX.X%) | 0.XXXX |
| Prone position | XXX : XXX (XXX.X%) | 0.XXXX |
| . Days with Mechanical Ventilation [days] | | TW |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Mean (SD) | XXX (XXX) | |
| Median (IQR) | XXX (XXX) | |

XXX~XXX

XXX~XXX

Prior Procedure: procedures onset prior to Day 1

O1~O3

Min~Max

Concomitant Procedures: procedures from Day 1 to End of Treatment Visit Post Procedure: procedures after End of Treatment Visit to End of Study Day# = End date/time - Start date/time, rounded up to the nearest integer



Protocol No.: CX4945-AV01-IIT

#### **Statistical Analysis Plan: Mock-up Tables and Figures**

Silmitasertib (CX-4945) for COVID-19

#### 14.1.9 Study Drug Administration, Compliance and Exposure

| Population: Intent-to-Treat Population | and Exposure |
|---|---|
| Characteristics | CX-4945 |
| . Repeat Variable: | |
| Treatment Duration [days], | |
| Total CX-4945 Dose [caps], | |
| Mean Daily Dose [caps / day] | |
| Total CX-4945 Administration [Times], | |
| Treatment Compliance [%], Mean Daily Administration [times / day] | |
| N (Missing) | XXX |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| . Treatment Compliance | |
| N (Missing) | XXX (XXX) |
| <50% | XXX (XXX.X%) |
| 50 ~ <75% | XXX (XXX.X%) |
| 75 ~ <100% | XXX (XXX.X%) |
| 100 ~ <125% | XXX (XXX.X%) |
| ≥125% | XXX (XXX.X%) |
| . CX-4945 Completion | |
| N | XXX |
| CX-4945 Completed | XXX (XXX.X%) |
| CX-4945 Not Completed | XXX (XXX.X%) |
| ~ Drug Interruption | XXX (XXX.X%) |
| ~ Drug Discontinuation | XXX (XXX.X%) |
| ~ <reason 1=""></reason> | XXX (XXX.X%) |
| ~ <reason 2=""></reason> | XXX (XXX.X%) |
| | ( - , -) |

Treatment Duration [days] = the last administration date – the first administration + Adjustment

| The first administration time | The last administration time | Adjustment |
|-------------------------------|------------------------------|------------|
| Morning | Morning | +0.5 |
| Morning | Evening | +1 |
| Evening | Morning | +0 |
| Evening | Evening | +0.5 |

Mean Daily Dose [caps / day] = Total CX-4945 Dose [caps] / Treatment Duration [days]

# of times of CX-4945 actually administered Treatment Compliance [%]=

(Treatment Duration) \* (2 times of administration/day)

Mean Daily Administration [times / day] = Total CX-4945 Administration [Times] / Treatment Duration [days]

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc.

Silmitasertib (CX-4945) for COVID-19

#### 14.2 EFFICACY DATA

#### <TTR Layout: For Time to Response Data>

Population: Intent-to-Treat Population / Per-Protocol Population

| Characteristics Treatment Group Difference P-value |
|----------------------------------------------------|
|----------------------------------------------------|

--Repeat Population: <See populations above>

#### - Variable per table title:

Time to COVID-19-Related Clinical Signs Normalization [days]

Time to COVID-19-Related Symptoms Resolution [days]

Time to SARS-COV-2 Viral Clearance [days]

#### . Repeat Scenario: Best Case Scenario, Worst Case Scenario

| N (Missing) | XXX (XXX) | LOGRANK |
|-----------------|-------------|---------|
| Censored No. | XXX (XXX%) | 0.XXXX |
| Observed No. | XXX (XXX%) | |
| Q1 [95% CI] | XXX [XX~XX] | |
| Median [95% CI] | XXX [XX~XX] | |
| Q3 [95% CI] | XXX [XX~XX] | |
| Mean (SE) | XXX (XXX) | |
| Min | XXX | |
| Max (Observed) | XXX | |
| Max | XXX | |

Footnote the definition according to [Instructions and Abbreviations] of title pages.

#### <TTR Figure Layout: For Response Proportion>





Silmitasertib (CX-4945) for COVID-19

#### 14.2.1 **COVID-19-Related Clinical Signs**

Time to COVID-19-Related Clinical Signs Normalization 14.2.1.1

Use TTR Layout

Footnote: refer to table 14.3.8 for the normal status of each symptom by visit

- 14.2.1.2 Figure of Normalization Proportion on COVID-19-Related Clinical Signs (Best Case Scenario)
- Figure of Normalization Proportion on COVID-19-Related Clinical Signs 14.2.1.3 (Worst Case Scenario)

Use TTR Figure Layout

- 14.2.1.4 **Time to Oxygen Saturation Level Normalization** Use TTR Layout
  - 14.2.1.5 Figure of Normalization Proportion on Oxygen Saturation Level (Best Case Scenario)
  - 14.2.1.6 Figure of Normalization Proportion on Oxygen Saturation Level (Worst **Case Scenario**)

Use TTR Figure Layout

#### **Covid-19-Related Symptoms** 14.2.2

- 14.2.2.1 Time to COVID-19-Related Symptoms Resolution Use TTR Layout
  - 14.2.2.2 Figure of Recovery Proportion on COVID-19-Related Symptoms (Best Case Scenario)
  - Figure of Recovery Proportion on COVID-19-Related Symptoms (Worst 14.2.2.3 Case Scenario)

Use TTR Figure Layout

Version 1.0, 25-JAN-2022 Protocol No.: CX4945-AV01-IIT



Silmitasertib (CX-4945) for COVID-19

#### 14.2.3 Nasopharyngeal Swab RT-PCR Result and SARS-COV-2 Viral Load

#### 14.2.3.1 SARS-COV-2 Viral Clearance and Viral Load [copies/µL]

| Population: | Intent-to-Treat Pop | ulation / | Per-Protocol | Pop | ulation |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

Treatment Group Difference P-value Characteristics --Repeat Population: <See populations above> . Repeat Visit: Visit 1 (Screening), Baseline, Visit 4 (Day 8), Visit 6 (Day 14, EOT), Visit 7 (Day 28, F1), LOCF N (Missing) XXX (XXX) Negative XXX (XXX.X%) Positive XXX (XXX.X%) N (Missing) XXX (XXX) 0.XXXXMean (SD) XXX (XXX) Median (IQR) XXX (XXX) Q1~Q3 XXX~XXX Min~Max XXX~XXX Repeat [Baseline to Visit] except Visit 1 (Screening) and Baseline C/F N (Missing) XXX (XXX) 0.XXXX Positive to Negative# XXX (XX.X%) Positive to Positive XXX (XX.X%) Diff. between groups §C - §S Difference (#) XXX% 95% CI (#) XXX%~XXX%a Repeat [Visit - Baseline] except Visit 1 (Screening) and Baseline TWN (Missing) XXX (XXX) 0.XXXXMean (SD) XXX (XXX) Median (IQR) XXX (XXX) Q1~Q3 XXX~XXX Min~Max XXX~XXX For W, normality is not applied Groups Diff §C - §S Median (Asymptotic SE) XXX95% CI (HL) XXX~XXX For T, normality is applied Groups Diff §C - §S Mean (SD) XXX (XXX) 95% CI XXX~XXX

a denotes CI using normal approximation for binomial proportion of # Viral Load > 25,000.00 copies/ $\mu$ L is estimated as 25,000.00 copies/ $\mu$ L. Baseline is Visit 2 (Day 1) data, or is Visit 1 if Visit 2 (Day 1) is null

Time to SARS-COV-2 Viral Clearance 14.2.3.2

Use TTR Layout

Figure of SARS-COV-2 Viral Clearance Proportion (Best Case Scenario) 14.2.3.3

14.2.3.4 Figure of SARS-COV-2 Viral Clearance Proportion (Worst Case Scenario)

Use TTR Figure Layout

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc. Protocol No.: CX4945-AV01-IIT A2 Healthcare Taiwan Co. 



Silmitasertib (CX-4945) for COVID-19

# 14.2.4 Clinical Status - NIAID 8-Point Clinical Progression Outcomes Scale

#### 14.2.4.1 Clinical Status - NIAID 8-Point Clinical Progression Outcomes Scale

Population: Intent-to-Treat Population / Per-Protocol Population

| Characteristics | Treatment Group | • | P-value |
|---|---|---|---|
| Repeat Population: <see above="" populations=""></see> | | | |
| N Subjects with any below [Event#:Subj#] ~ Death (NIAID item 1) ~ Respiratory Failure (NIAID item 2~3 or from AE) ~ Hospitalized (NIAID item 2~6) | XXX<br>XXX: XXX (XXX.X%)<br>XXX: XXX (XXX.X%)<br>XXX: XXX (XXX.X%)<br>XXX: XXX (XXX.X%) | | |
| . Repeat Visit: No 'Visit 1 (Screening)' for IL-6:<br>Visit 1 (Screening), Baseline,<br>Adjusted Visit 3 (Day 4), Adjusted Visit 4 (Day 8), | | | |
| Adjusted Visit 5 (Day 11), Adjusted Visit 6 (Day 14, EOT Visit 7 (Day 28, F1), Visit 8 (Day 45, F2), LOCF | Γ), | | |
| | XXX (XXX) XXX (XXX.X%) XXX (XXX.X%) | | 0.XXXX |
| Visit 7 (Day 28, F1), Visit 8 (Day 45, F2), LOCF N (Missing) Item 1 | XXX (XXX)<br>XXX (XXX.X%) | | 0.XXXX |

Respiratory failure required mechanical ventilation, oxygen delivered by high-flow nasal cannula, ESMO; shock or multi-organ dysfunction/failure

XXX (XX.X%)

X

For NIAID 8-Point Clinical Progression Outcomes Scale:

Item 1 - Death

Item 2~3 - Hospitalized, respiratory failure

Progression (Item 7 to Item 1~6)

Item 4~6 - Hospitalized, non-respiratory failure

Item 7 - Not hospitalized, limitation on activities and/or requiring home oxygen

Item 8 - Not hospitalized, no limitations on activities

Refer to [Instructions and Abbreviations] of title pages for further definition

# 14.2.4.2 Time to Improvement on NIAID 8-Point Clinical Progression Outcomes Scale

Use TTR Layout

# 14.2.4.3 Figure of Improvement Proportion on NIAID 8-Point Clinical Progression Outcomes Scale (Best Case Scenario)

# 14.2.4.4 Figure of Improvement Proportion on NIAID 8-Point Clinical Progression Outcomes Scale (Worst Case Scenario)

Use TTR Figure Layout

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc. Protocol No.: CX4945-AV01-IIT  A2 Healthcare Taiwan Co.



Silmitasertib (CX-4945) for COVID-19

#### 14.2.5 EQ-5D-5L

#### 14.2.5.1 EQ-5D-5L

| Population: I | Intent-to-Treat P | opulation / | Per-Protocol | Population |
|---------------|-------------------|-------------|--------------|------------|
|---------------|-------------------|-------------|--------------|------------|

| Characteristics | Treatment Group | Difference | P-value |
|---|---|---|---|
| Repeat Population: <see above="" populations=""></see> | 1 | | |
| Repeat Visit: | EOE) III : I T (D 20 | E1) LOGE | |
| Visit 2 (Day 1), Visit 4 (Day 8), Visit 6 (Day 14, F | 201), Visit / (Day 28, | F1), LOCF | |
| . Repeat Variable: | | | TW |
| Total score of Q1~Q5, Imaginable Health Status | | | (Visit 2 (Day 1)) |
| N (Missing) | XXX (XXX) | | 0.XXXX |
| Mean (SD) | XXX (XXX) | | |
| Median (IQR) | XXX (XXX) | | |
| Q1~Q3 | XXX~XXX | | |
| Min~Max | XXX~XXX | | |
| For Imaginable Health Status only | | | |
| > 90 | XXX (XXX.X%) | | |
| < 90 | XXX (XXX.X%) | | |
| Repeat [Visit - Visit 2 (Day 1)] except Visit 2 (Day | , | | |
| N (Missing) | XXX (XXX) | | TW |
| N (Missing) | XXX (XXX) | | 0.XXXX |
| Mean (SD) | XXX(XXX) | | |
| Median (IQR) | XXX(XXX) | | |
| Q1~Q3 | XXX~XXX | | |
| Min~Max | XXX~XXX | | |
| For W, normality is not applied | | §C - §S | |
| Groups Diff | | 0 - 0 - | |
| Median (Asymptotic SE) | | XXX | |
| 95% CI (HL) | | XXX~XXX | |
| For T, normality is applied | | §C - §S | |
| Groups Diff | | | |
| Mean (SD) | | XXX (XXX) | |
| 95% CI | | XXX~XXX | |

Q1. Mobility, Q2. Self-Care, Q3. Usual Activities, Q4. Pain/Discomfort, Q5. Anxiety/Depression

# 14.2.5.2 Time to Improvement on EQ-5D-5L Imaginable Health Status Use TTR Layout

# 14.2.5.3 Figure of Improvement Proportion on EQ-5D-5L Imaginable Health Status (Best Case Scenario)

# 14.2.5.4 Figure of Improvement Proportion on EQ-5D-5L Imaginable Health Status (Worst Case Scenario)

Use TTR Figure Layout

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc. Protocol No.: CX4945-AV01-IIT  A2 Healthcare Taiwan Co.



Silmitasertib (CX-4945) for COVID-19

#### 14.3 SAFETY DATA

#### 14.3.1 Treatment Emergent Adverse Event – Subject Based Analyses

#### 14.3.1.1 Treatment Emergent AE - Summary

Population: Safety Population

| Characteristics [Event#:Subj#] | Treatment Group |
|---------------------------------------------|--------------------|
| (Multi-Selection) | |
| N | XXX |
| Subjects with AE | XXX: XXX (XXX.X%) |
| ~ Grade ≥3 | XXX : XXX (XXX.X%) |
| ~ Grade 4 | XXX : XXX (XXX.X%) |
| ~ Grade 5 | XXX : XXX (XXX.X%) |
| Subjects with Treatment-Related AE | XXX: XXX (XXX.X%) |
| ~ Grade ≥3 | XXX : XXX (XXX.X%) |
| ~ Grade 4 | XXX : XXX (XXX.X%) |
| ~ Grade 5 | XXX : XXX (XXX.X%) |
| Subjects with AE Leading to Action Taken | XXX: XXX (XXX.X%) |
| ~ Dose Reduced | XXX: XXX (XXX.X%) |
| ~ Drug Interrupted | XXX : XXX (XXX.X%) |
| ~ Drug Withdrawn by Subject | XXX : XXX (XXX.X%) |
| ~ Drug Withdrawn Instructed by Investigator | XXX : XXX (XXX.X%) |
| Subjects with SAE | XXX : XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX: XXX (XXX.X%) |
| ~ Life-Threatening SAE | XXX: XXX (XXX.X%) |
| ~ Death SAE | XXX:XXX(XXX.X%) |
| ~ SUSAR | XXX: XXX (XXX.X%) |
| ~ Death SUSAR | XXX: XXX (XXX.X%) |

Subject with multiple events are counted as one incidence.

Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related

#### 14.3.1.2 Treatment Emergent AE - Subjects with AE

#### 14.3.1.3 Treatment Emergent AE - Subjects with Treatment-Related AE

Population: Safety Population

| Characteristics | Treatment Group |
|---|---|
| (Multi-Selection by XXX, System Organ Class and Preferred Term) | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX : XXX (XXX.X%) |
| ~ <meddra body="" system1=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Body System2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX : XXX (XXX.X%) |

For each MedDRA (version 23.1) SOC or Preferred Term, subject with multiple events are counted as one incidence.

[For 14.3.1.3] Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc. Protocol No.: CX4945-AV01-IIT  A2 Healthcare Taiwan Co.



Silmitasertib (CX-4945) for COVID-19

#### 14.3.1.4 Treatment Emergent AE - Subjects with Grade ≥3 AE

#### 14.3.1.5 Treatment Emergent AE - Subjects with Grade ≥3 Treatment-Related AE

Population: Safety Population

| Characteristics | Treatment Group |
|---|---|
| (Multi-Selection by Severity Grade, System Organ Class and Preferred Term) | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| ~ Repeat Severity Grade: | |
| Grade ≥3, Grade 4, Grade 5 | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System2> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX:XXX(XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |

[For 14.3.1.5] Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related

#### 14.3.1.6 Treatment Emergent AE - Subjects with AE Leading to Action Taken

Population: Safety Population

| Characteristics | Treatment Group |
|---|---|
| (Multi-Selection by Action Taken, System Organ Class and Preferred Term) | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX : XXX (XXX.X%) |
| ~ Repeat Action Taken: | |
| Dose Increased, Dose Reduced, Drug Interrupted, | |
| Drug Withdrawn by Subject, | |
| Drug Withdrawn Instructed by Investigator | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System1> | XXX:XXX(XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX:XXX(XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |



Silmitasertib (CX-4945) for COVID-19

#### 14.3.1.7 Treatment Emergent AE – Subjects with Serious Adverse Event (SAE)

# 14.3.1.8 Treatment Emergent AE – Subjects with Suspected Unexpected Serious Adverse Reaction (SUSAR)

SUSAR: Unexpected Treatment Related SAE

Population: Safety Population

| Characteristics | Treatment Group |
|---|---|
| (Multi-Selection by SAE Criteria, System Organ Class | s and Preferred Term) |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| Repeat SAE Criterion: | |
| Any SAE Criterion, Requires or Prolongs Hospitalizat | tion, |
| death, | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |

SAE Criteria 'F/L/H' and 'F/L' will be counted as 'F' only, and 'L/H' as 'L', where F=Fatal (Death), L=Life threatening, H=Require hospitalization or prolongation of existing hospitalization.



Silmitasertib (CX-4945) for COVID-19

| 14.3.2 | Laboratory | <b>Examination</b> | <ul> <li>Hematology</li> </ul> |
|--------|------------|--------------------|--------------------------------|

- 14.3.2.1 Hematology <Item 1 and Unit>
- 14.3.2.2 Hematology <Item 2 and Unit>
- 14.3.2.3 .... Refer to [Instructions and Abbreviations] of section 16 for the test terms

#### 14.3.3 Laboratory Examination – Chemistry

- 14.3.3.1 Chemistry <Item 1 and Unit>
- 14.3.3.2 Chemistry <Item 2 and Unit>
- 14.3.3.3 .... Refer to [Instructions and Abbreviations] of section 16 for the test terms

#### 14.3.4 Laboratory Examination – Inflammatory Marker

- 14.3.4.1 Inflammatory Marker <Item 1 and Unit>
- 14.3.4.2 Inflammatory Marker <Item 2 and Unit>
- 14.3.4.3 .... Refer to [Instructions and Abbreviations] of section 16 for the test terms

#### 14.3.5 Laboratory Examination – Coagulation

- 14.3.5.1 Coagulation <Item 1 and Unit>
- 14.3.5.2 Coagulation <Item 2 and Unit>
- 14.3.5.3 .... Refer to [Instructions and Abbreviations] of section 16 for the test terms

#### 14.3.6 Laboratory Examination – Urinalysis

- 14.3.6.1 Urinalysis <Item 1 and Unit>
- 14.3.6.2 Urinalysis <Item 2 and Unit>
- 14.3.6.3 .... Refer to [Instructions and Abbreviations] of section 16 for the test terms

# <LB Layout 1: For Continuous Laboratory Test; Clinical relevance analyses will be excluded if not applicable>

Population: Safety Population

| Characteristics | Treatment Group | Difference | p-value |
|---|---|---|---|
| . Repeat Visit: No 'Visit 1 (Screening)' for IL-6: | | | |
| Visit 1 (Screening), Baseline, | | | |
| Adjusted Visit 3 (Day 4), Adjusted Visit 4 (Day 8), | | | |
| Adjusted Visit 5 (Day 11), Adjusted Visit 6 (Day 14 | , EOT), | | |
| Visit 7 (Day 28, F1), Visit 8 (Day 45, F2) | | | T/W |
| | | | <baseline only=""></baseline> |
| N (Missing) | XXX (XXX) | | 0.XXXX |
| Mean (SD) | XXX (XXX) | | |
| Median (IQR) | XXX (XXX) | | |
| Q1~Q3 | $XXX\sim XXX$ | | |
| Min~Max | $XXX\sim XXX$ | | |
| For W, normality is not applied <baseline only=""></baseline> | | | |
| Groups Diff | | §C - §S | |
| Median (Asymptotic SE) | | XXX | |
| 95% CI (HL) | | $XXX\sim XXX$ | |



Silmitasertib (CX-4945) for COVID-19

| Characteristics | Treatment Group | Difference | p-value |
|---|---|---|---|
| For T, normality is applied <baseline only=""></baseline> | | | |
| Groups Diff | | §C - §S | |
| Mean (SD) | | XXX (XXX) | |
| 95% CI | | XXX~XXX | |
| N (Missing) | XXX (XXX) | | |
| Normal | XXX (XX.X%) | | |
| NCS | XXX (XX.X%) | | |
| CS (Medical History) | XXX (XX.X%) | | |
| CS (Adverse Event) | XXX (XX.X%) | | |
| | 11111 (11111170) | | |
| . Repeat [Visit – Baseline] excluding Visit 1 (Screen | ing) and Baseline | | ANCOVA/W |
| N (Missing) | XXX (XXX) | | 0.XXXX |
| Mean (SD) | XXX (XXX) | | |
| Median (IQR) | XXX (XXX) | | |
| Q1~Q3 | XXX~XXX | | |
| Min~Max | $XXX\sim XXX$ | | |
| 95% CI (WI) | XXX~XXXwt | | |
| For W, normality is not applied | | | |
| Groups Diff | | §C - §S | |
| 95% CI (HL) | | XXX~XXX | |
| For ANOVA, normality is applied | XXX (XXX) | | |
| LsMean (SE) | XXX~XXX | | |
| 95% CI of LsMean | | | |
| Groups Diff. (T) | | §C- §S | |
| Difference of LsMean | | XXX | |
| 95% CI of LsMean | | XXX~XXX | |
| | | <b></b> | |

ANCOVA Model (p-value 0.XXXX) with effect Treatment (p-value 0.XXXX), Baseline (p-value 0.XXXX), Treatment\*Baseline (p-value 0.XXXX).

| . Repeat | [ <baseline> to <visit>]</visit></baseline> |
|----------|---------------------------------------------|
| NT /N f | . \ |

Protocol No.: CX4945-AV01-IIT

| N (Missing) | XXX (XXX) |
|----------------------------|-------------|
| Relieved | XXX (XX.X%) |
| Unchanged | XXX (XX.X%) |
| Worsened (Medical History) | XXX (XX.X%) |
| Worsened (Adverse Event) | XXX (XX.X%) |

For Item excluding IL-6 Baseline is Visit 2 (Day 1) data, or is Visit 1 if Visit 2 (Day 1) is null For IL-6 Baseline is Visit 2 (Day 1) data

Refer to [Instructions and Abbreviations] of title pages for Transition of Clinical Relevance

A2 Healthcare Taiwan Co.



# <LB Layout 2: For Categorical Urinalysis Test, including pH;</p> MHCHISQ for PH, C/F for else>

Population: Safety Population

| Characteristics | Transment Comme | n |
|---|---|---|
| Characteristics Percet Visit: | Treatment Group | p-value |
| Repeat Visit: | | |
| Visit 1 (Screening), Baseline, | | |
| Adjusted Visit 3 (Day 4), Adjusted Visit 4 (Day 8), | | |
| Adjusted Visit 5 (Day 11), Adjusted Visit 6 (Day 14, EOT), | | MHCHISQ / |
| Visit 7 (Day 28, F1), Visit 8 (Day 45, F2) | | C/F |
| NI (Mississe) | VVV (VVV) | <baseline only=""></baseline> |
| N (Missing) | XXX (XXX) | 0.XXXX |
| <value 1=""></value> | XXX (XX.X%) | |
| <value 2=""></value> | XXX (XX.X%) | |
| <value 3=""></value> | XXX (XX.X%) | |
| N (Missing) | XXX (XXX) | |
| Normal | XXX (XX.X%) | |
| NCS | XXX (XX.X%) | |
| CS (Medical History) | XXX (XX.X%) | |
| CS (Adverse Event) | XXX (XX.X%) | |
| . Repeat [ <visit> - <baseline>] for pH</baseline></visit> | | |
| Repeat [ <baseline> to <visit>] for else</visit></baseline> | | MHCHISQ / |
| For <visit> excluding Visit 1 (Screening) and Baseline</visit> | | C/F |
| N (Missing) | XXX (XXX) | 0.XXXX |
| <value 1=""></value> | XXX (XX.X%) | |
| <value 2=""></value> | XXX (XX.X%) | |
| <value 3=""></value> | XXX (XX.X%) | |
| | , , , | |
| . Repeat [ <baseline> to <visit>]</visit></baseline> | | |
| N (Missing) | XXX(XXX) | |
| Relieved | XXX (XX.X%) | |
| Unchanged | XXX (XX.X%) | |
| Worsened (Medical History) | XXX (XX.X%) | |
| Worsened (Adverse Event) | XXX (XX.X%) | |

Baseline is Visit 2 (Day 1) data, or is Visit 1 if Visit 2 (Day 1) is null

Refer to [Instructions and Abbreviations] of title pages for Transition of Clinical Relevance

[For Color and Appearance] Data of normal values will be coded as 'Normal', and data not in normal values will be coded as 'Abnormal'.



Silmitasertib (CX-4945) for COVID-19

#### 14.3.7 Physical Examination

#### 14.3.7.1 Physical Examination – All Abnormalities

Population: Safety Population

| Characteristics | Treatment Group |
|---|---|
| . Repeat Visit: | |
| Visit 1 (Screening), Visit 2 (Day 1), Visit 4 (Day 8), | |
| Visit 6 (Day 14, EOT), Visit 7 (Day 28, F1), Visit 8 (Day 45, F2) | |
| N (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ NCS | XXX (XXX.X%) |
| ~CS (Medical History) | XXX (XXX.X%) |
| ~CS (Adverse Event) | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ NCS | XXX (XXX.X%) |
| ~CS (Medical History) | XXX (XXX.X%) |
| ~CS (Adverse Event) | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ NCS | XXX (XXX.X%) |
| ~CS (Medical History) | XXX (XXX.X%) |
| ~CS (Adverse Event) | XXX (XXX.X%) |
| ••• | ••• |

#### 14.3.8 Vital Signs, Body Weight and SpO2

| 14.3.8.1 | vitai Signs – Temperature [degree C] |
|----------|----------------------------------------------|
| 14.3.8.2 | Vital Signs – Respiratory Rate [breaths/min] |
| 14.3.8.3 | Vital Signs – Systolic Blood Pressure [mmHg] |
| 11201 | THE ICE OF A PERSON OF THE |

14.3.8.4 Vital Signs – Diastolic Blood Pressure [mmHg]

14.3.8.5 Vital Signs – Heart Rate [beats/min]

14.3.8.6 Vital Signs – Weight [kg]

14.3.8.7 Vital Signs – Pulse Oxygen Saturation (SpO2) [%]



Silmitasertib (CX-4945) for COVID-19

| Population: Safety Population | | |
|---|---|---|
| Characteristics | Treatment Group | p-value |
| . Repeat Visit: | | |
| Visit 1 (Screening), Baseline, | | |
| Adjusted Visit 3 (Day 4), Adjusted Visit 4 (Day 8), Adjusted Visit 4 (Day 8), Adjusted Visit 4 (Day 8), Adjusted Visit 5 (Day 8), Adjusted Visit 5 (Day 8), Adjusted Visit 6 (Day 8), Adjusted Visit 6 (Day 8), Adjusted Visit 7 (Day 8), Adjusted Visit 8 (Day 8), Adjusted Visit 9 ( | usted Visit 5 (Day 11), | T/W |
| Adjusted Visit 6 (Day 14, EOT), Visit 7 (Day 28, F1), V | visit 8 (Day 45, F2) | <baseline only=""></baseline> |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Mean (SD) | XXX (XXX) | |
| Median (IQR) | XXX (XXX) | |
| Q1~Q3 | XXX~XXX | |
| Min~Max | XXX~XXX | |
| For W, normality is not applied | §C - §S | |
| Groups Diff | | |
| Median (Asymptotic SE) | XXX | |
| 95% CI (HL) | XXX~XXX | |
| | 12.2.2 | |
| For T, normality is applied | §C - §S | |
| Groups Diff | 2C 2D | |
| Mean (SD) | XXX (XXX) | |
| 95% CI | XXX~XXX | |
| 75,70 5- | MM MM | |
| For Temperature, Respiratory Rate, Heart Rate, | | |
| Pulse Oxygen Saturation (SpO2) | | C/F |
| Normal | XXX (XXX.X%) | 0.XXXX |
| Abnormal | XXX (XXX.X%) | V |
| | ( | |
| . Repeat [Visit – Baseline] excluding Visit 1 (Screening) | ANCOVA/W | |
| N (Missing) | XXX (XXX) | 0.XXXX |
| Mean (SD) | XXX (XXX) | |
| Median (IQR) | XXX (XXX) | |
| Q1~Q3 | XXX~XXX | |
| Min~Max | XXX~XXX | |
| 95% CI (WI) | XXX~XXXwt | |
| For W, normality is not applied | <\$C - \$S> | |
| Groups Diff | XXX~XXX | |
| 95% CI (HL) | AAA -AAA | |
| For ANCOVA, normality is applied | XXX (XXX) | |
| <i>y</i> 3 11 | XXX~XXX | |
| LsMean (SE) | | |
| 95% CI of LsMean | | |
| Groups Diff. (T) | <\$C- \$S> | |
| Difference of LsMean | XXX | |
| 95% CI of LsMean | XXX~XXX | |
| • | AAA~AAA | |
| ANGOVA M. 1-1 (1 0 VVVV) - 14- CC4 To4- | ( 1 0 XXXXX) D 1' | ( 1 |

ANCOVA Model (p-value 0.XXXX) with effect Treatment (p-value 0.XXXX), Baseline (p-value 0.XXXX), Treatment\*Baseline (p-value 0.XXXX).

Baseline is Visit 2 (Day 1) data, or is Visit 1 if Visit 2 (Day 1) is null

[Temperature] Normal: <36.6°C from axillary site, or < 37.2°C from oral site or < 37.8°C from rectal or tympanic site

[Respiratory Rate] Normal: < 20 breaths/min

[Heart Rate] Normal: <90 beats/min

[Pulse Oxygen Saturation (SpO2)] Normal: ≥ 96%

Version 1.0, 25-JAN-2022 Confidential Senhwa Biosciences, Inc. A2 Healthcare Taiwan Co. Protocol No.: CX4945-AV01-IIT 



#### Electrocardiogram (ECG) 14.3.9

#### **Electrocardiogram - Overall interpretation** 14.3.9.1

Population: Safety Population

| Characteristics | Treatment Group |
|------------------------------------------------|-----------------|
| . Visit 1 (Screening), Visit 6 (Day 14, EOT), | |
| N (Missing) | XXX (XXX) |
| Normal | XXX(XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| . Visit 1 (Screening) to Visit 6 (Day 14, EOT) | |
| N (Missing) | XXX (XXX) |
| Relieved | XXX(XX.X%) |
| Unchanged | XXX(XX.X%) |
| Worsened (Medical History) | XXX (XX.X%) |
| Worsened (Adverse Event) | XXX (XX.X%) |

Version 1.0, 25-JAN-2022 Protocol No.: CX4945-AV01-IIT